CLINICAL TRIAL: NCT03252613
Title: Translational Approaches to Septic Cardiomyopathy
Acronym: TASC01
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samuel Brown (Other)
Collaborators: Euan Ashley (Unknown)
Responsible Party: Sponsor-Investigator, Samuel Brown, Principal Investigator, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Other Study IDs: 1050374
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Cardiomyopathies; Sepsis; Septic Shock
Keywords: septic cardiomyopathy; cytokine; iPSC; Inducible pluripotent stem cell
MeSH Terms: conditions — Cardiomyopathies; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This translational study will assess the association between septic cardiomyopathy (measured via left ventricular global longitudinal strain) and (a) inflammatory cytokine profiles, and (b) the behavior of cardiomyocytes derived from inducible pluripotent stem cells.

ELIGIBILITY:
INCLUSION CRITERIA

At least 18 years of age Admitted to the ICU

SEPSIS PATIENTS:

Sepsis patients must have:

1. Suspected or confirmed infection AND
2. Organ dysfunction as defined by a SOFA >= 2 above baseline (if no baseline data available, SOFA assumed to be 0)

OR

SEPTIC SHOCK PATIENTS:

AFTER INFUSION OF 20ML/KG CRYSTALLOID OR EQUIVALENT, septic shock patients must have:

1. Suspected or confirmed infection AND
2. Lactate > 2 mmol/L AND
3. Receiving vasopressors

EXCLUSION CRITERIA Known pregnancy Primary diagnosis of acute coronary syndrome Known preexisting heart disease Known severe valvular disease (regurgitation or stenosis)

Major cardiac dysrhythmia such as:

* Ventricular tachycardia (V-tach)
* Ventricular Fibrillation (V-fib)
* Third degree heart block (complete hear block or complete AV block)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of study subjects must be 18 years of age, admitted to an ICU and have sepsis or septic shock as defined in the above inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-10-27 (Estimated); Study Completion 2019-10-27 (Estimated)

PRIMARY OUTCOMES:
Correlation of cytokine profile with left ventricular global longitudinal strain | Day 1
  This outcome assesses the correlation between inflammatory cytokines (summarized via PCA) and septic cardiomyopathy, as assessed by left ventricular global longitudinal strain.

SECONDARY OUTCOMES:
Adrenergic susceptibility of pluripotent stem cell-derived cardiomyocytes | Day 1
  This is a laboratory-based outcome, using pluripotent stem cell-derived cardiomyocytes, with exposure to adrenergic agonists and antagonists in vitro

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, MD, Principal Investigator — Intermountain Health Care, Inc.; Euan Ashley, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Intermoutain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
There will be a database/tissue bank for future research